CLINICAL TRIAL: NCT01472003
Title: An Evaluation of the Biodistribution and Imaging Characteristics of ABT-806i (111In-ABT-806) in Subjects With Advanced Solid Tumor Types Likely to Express Epidermal Growth Factor Receptor (EGFR)
Brief Title: An Evaluation of the Biodistribution and Imaging Characteristics of ABT-806i (111In-ABT-806) in Subjects With Advanced Solid Tumor Types
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M11-849
Record Dates: First submitted 2011-10-12; First posted 2011-11-16 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — depatuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-806 Arm (Experimental): Subjects with advanced solid tumors
  Interventions: Drug: ABT-806
- ABT-806i Arm (Experimental): Subjects with advanced solid tumors
  Interventions: Drug: ABT-806i

INTERVENTIONS:
Drug: ABT-806 — ABT-806 will be administered by intravenous infusion.
  Arms: ABT-806 Arm
Drug: ABT-806i — ABT-806i will be administered by intravenous infusion.
  Arms: ABT-806i Arm

SUMMARY:
This is an open label study designed to evaluate the biodistribution and imaging characteristics of ABT-806i (111In-ABT-806) in subjects with advanced solid tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a solid tumor of a type likely or known to either overexpress wild-type Epidermal Growth Factor Receptor (EGFR) or to express variant III mutant EGFR (e.g., head and neck squamous cell carcinoma, Non-small Cell Lung Carcinoma (NSCLC), and colorectal carcinoma).
* Subject must have disease that is not amenable to surgical resection or other approved therapeutic options with curative intent.
* Subject cannot tolerate or must not be eligible for other approved therapeutic options with known survival advantage.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Subject must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 with at least 1 extrahepatic 2 cm lesion.

Exclusion Criteria:

* Subject has received anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational therapy within a period of 14 days prior to the first dose of ABT-806i.
* Subject has received a prior EGFR-directed monoclonal antibody within a period of 4 weeks prior to the first dose of ABT-806i.
* Subject has unresolved clinically significant toxicities from prior anticancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher.
* Subject has had major surgery within 21 days prior to the first dose of ABT-806i.
* Subject has a clinically significant uncontrolled condition(s) including but not limited to the following:

  * Active uncontrolled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Single-Photon Emission Computerized Tomography (SPECT) | Week 1
  Tumor receptor occupancy (Cohort 1 and Cohort 2)
Single-Photon Emission Computerized Tomography (SPECT) | Week 6
  Tumor receptor occupancy (Cohort 2)
Whole body planar imaging | Week 1
  Biodistribution and dosimetry (Cohort 1 and Cohort 2)
Whole body planar imaging | Week 6
  Biodistribution and dosimetry (Cohort 2)

SECONDARY OUTCOMES:
Pharmacokinetic profile evaluation - Cohort 1 | From Day 1 through Final Visit
  Blood samples for ABT-806/ABT-806i will be collected and assayed at designated timepoints
Pharmacokinetic profile evaluation - Cohort 2 | From Day 1 through Final Visit
  Blood samples for ABT-806/ABT-806i will be collected and assayed at designated timepoints
Single-Photon Emission Computerized Tomography (SPECT) | Week 1
  ABT-806i uptake correlation with Epidermal Growth Factor Receptor (EGFR) vIII expression - Cohort 2
Single-Photon Emission Computerized Tomography (SPECT) | Week 6
  ABT-806i uptake correlation with EGFR vIII expression - Cohort 2
Whole body planar imaging | Week 1
  ABT-806i uptake correlation with Epidermal Growth Factor Receptor (EGFR) vIII expression - Cohort 2
Whole body planar imaging | Week 6
  ABT-806i uptake correlation with EGFR vIII expression - Cohort 2
Blood pressure - Cohort 1 | Screening through Week 2
Heart rate - Cohort 1 | Screening through Week 2
Body temperature - Cohort 1 | Screening through Week 2
Number of subjects with Adverse Events - Cohort 1 | Day 1 Through Week 2
  The investigator will monitor each subject for clinical and laboratory evidence of adverse events.
Chemistry - Cohort 1 | Sceening, Week 1 and Final Visit
Hematology - Cohort 1 | Sceening, Week 1 and Final Visit
Urinalysis - Cohort 1 | Sceening, Week 1 and Final Visit
Physical Examination - Cohort 1 | Screening, Week 1 and Final Visit
  Physical exam including body weight will be performed.
Electrocardiogram (ECG) - Cohort 1 | Baseline and Final Visit
  12-lead ECG will be performed.
Heart rate - Cohort 2 | Screening Through Week 8
Blood pressure - Cohort 2 | Screening Through Week 8
Number of subjects with Adverse Events - Cohort 2 | Day 1 Through Week 8
  The investigator will monitor each subject for clinical and laboratory evidence of adverse events.
Body temperature - Cohort 2 | Screening Through Week 8
Hematology - Cohort 2 | Screening, Week 1, 2, 4, 6, and Final Visit
Chemistry - Cohort 2 | Screening, Week 1, 2, 4, 6, and Final Visit
Physical Examination - Cohort 2 | Screening, Week 1, 2, 4, 6, and Final Visit
  Physical exam including body weight will be performed.
Urinalysis - Cohort 2 | Screening, Week 1, 2, 4, 6, and Final Visit
Electrocardiogram (ECG) - Cohort 2 | Baseline and Week 6
  12-lead ECG will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle D. Holen, MD, Study Director — AbbVie
Locations (2):
- Australia (2):
  - Site Reference ID/Investigator# 52203, Heidelberg
  - Site Reference ID/Investigator# 58242, Herston

REFERENCES:
- [Derived] Gan HK, Burge M, Solomon B, Lee ST, Holen KD, Zhang Y, Ciprotti M, Lee FT, Munasinghe W, Fischer J, Ansell P, Fox G, Xiong H, Reilly EB, Humerickhouse R, Scott AM. A Phase 1 and Biodistribution Study of ABT-806i, an 111In-Radiolabeled Conjugate of the Tumor-Specific Anti-EGFR Antibody ABT-806. J Nucl Med. 2021 Jun 1;62(6):787-794. doi: 10.2967/jnumed.120.253146. Epub 2021 Jan 28. PMID 33509972